CLINICAL TRIAL: NCT00725855
Title: A Single-Center, Double-Blind, Placebo-Controlled, Randomized Blocks Study Investigating the Effect of 4 Dosages (1 mg, 5 mg, 15 mg, 50 mg) of MEM 3454 on P50 Sensory Gating and Mismatch Negativity (MMN) in Patients With Schizophrenia
Brief Title: A Single-Center, Double-Blind (DB) Study of MEM 3454 on P50 Sensory Gating and Mismatch Negativity in Schizophrenia Patients
Acronym: P50
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Memory Pharmaceuticals (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Abdul Abdullah, MD, Project Medical Director, Memory Pharmaceuticals Corp.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MEM 3454-102
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2008-07-31 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; P50 Sensory Gating; Mismatched Negativity
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): 1 mg dose
  Interventions: Drug: MEM 3454
- 2 (Experimental): 5 mg dose
  Interventions: Drug: MEM 3454
- 3 (Experimental): 15 mg dose
  Interventions: Drug: MEM 3454
- 4 (Experimental): 50 mg dose
  Interventions: Drug: MEM 3454
- 5 (Placebo Comparator): Placebo dose
  Interventions: Drug: Placebo for MEM 3454

INTERVENTIONS:
Drug: MEM 3454 — 1 mg dose
  Arms: 1
Drug: MEM 3454 — 5 mg dose
  Arms: 2
Drug: MEM 3454 — 15 mg dose
  Arms: 3
Drug: MEM 3454 — 50 mg dose
  Arms: 4
Drug: Placebo for MEM 3454 — Placebo dose
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the effects of nicotinic alpha-7 MEM 3454 on P50 sensory gating in patients with Schizophrenia. The hypothesis is that MEM 3454 will normalize the P50 ratio.

Data produced in this study will provide useful information regarding the value of P50 as an efficacy biomarker, and provide evidence for the optimal dosing of MEM 3454 for additional P50 studies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female subjects between 18and 55 years of age.
* 2. Fluent in English, even if English is not the primary language.
* 3. Able to provide informed consent.
* 4. DSM IV-R primary diagnosis of schizophrenia (any subtype), assessed using a structured diagnostic interview (SCID CT).
* 5. Few or no extra-pyramidal symptoms(EPS)at screening,defined as SAS < 6.
* 6. Negative urine drug screen (UDS).
* 7. Negative cotinine test.
* 8. Clinically stable, as judged by the investigator, and in a non-acute phase for at least 12 weeks. At least one month on the same dose of antipsychotic medication.

Exclusion Criteria:

* Current risk of suicide, or history of suicidal behavior within the last 6 months.
* Hospitalized for psychiatric symptoms in the past 3 months.
* Other psychiatric diagnoses.
* Substance abuse/dependence (other than nicotine or caffeine) within the last 6 months according to the SCID-CT.
* Currently smoking, nicotine replacement therapy, smoking cessation medications or remedies, including Varenicline (Chantix).
* Any medical condition, as judged by the Investigator, which may interfere with the subjects' participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-03 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Determine the utility of P50 sensory gating as an efficacy biomarker for nicotinic alpha-7 agonist such as MEM 3454. | Pre-dosing and Day 1

SECONDARY OUTCOMES:
• Investigate the safety and tolerability of MEM 3454 compared with placebo | all time points
• Determine whether MMN correlates with P50. | Pre-dose and day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ann Olincy, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States

REFERENCES:
- [Background] Braff DL, Light GA, Swerdlow NR. Prepulse inhibition and P50 suppression are both deficient but not correlated in schizophrenia patients. Biol Psychiatry. 2007 May 15;61(10):1204-7. doi: 10.1016/j.biopsych.2006.08.015. Epub 2006 Dec 8. PMID 17161386
- [Background] Olincy A, Harris JG, Johnson LL, Pender V, Kongs S, Allensworth D, Ellis J, Zerbe GO, Leonard S, Stevens KE, Stevens JO, Martin L, Adler LE, Soti F, Kem WR, Freedman R. Proof-of-concept trial of an alpha7 nicotinic agonist in schizophrenia. Arch Gen Psychiatry. 2006 Jun;63(6):630-8. doi: 10.1001/archpsyc.63.6.630. PMID 16754836
- [Background] Simosky JK, Stevens KE, Freedman R. Nicotinic agonists and psychosis. Curr Drug Targets CNS Neurol Disord. 2002 Apr;1(2):149-62. doi: 10.2174/1568007024606168. PMID 12769624